CLINICAL TRIAL: NCT00232713
Title: Uterine Fibroid Pregnancy Registry
Status: Terminated | Type: Observational
Sponsor: Syneos Health (Other)
Other Study IDs: AFB04-101
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Birth Defects; Pregnancy; Uterine Fibroids
Keywords: Birth Defects; Pregnancy; Uterine Fibroids; Fibroids
MeSH Terms: conditions — Congenital Abnormalities; Leiomyoma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The Uterine Fibroid Pregnancy Registry is a USA and European-based registry designed to monitor pregnancies in women with uterine fibroids in order to

1. estimate the risk ratio of birth defects in women with uterine fibroids who were treated or untreated during pregnancy and
2. detect any pattern of birth defects among pregnancies in specific treatment groups.

Those pregnant women exposed to various therapies used to treat uterine fibroids will be compared with those not exposed to treatment in order to detect any potential increase in the risk of major birth defects.

DETAILED DESCRIPTION:
This is a prospective, observational, registration and follow-up study of patients with uterine fibroids who become pregnant and their offspring. Those who are exposed to treatment at any time during pregnancy or within one month of conception will be compared with those not exposed to treatment. Enrollment of patients into the Registry may be initiated by health care providers and/or pregnant patients. Health care providers provide all information related to the pregnancy and the outcome.

During the study, data will be collected on uterine fibroids, exposure to treatment for uterine fibroids, potential confounding factors, and pregnancy outcome. Reported cases will be reviewed and classified according to type of birth defects. Registry enrollment is voluntary and should occur as early in pregnancy as possible, preferably before any prenatal testing. Midway between enrollment and the expected date of delivery, the Registry conducts a short interim follow-up with the health care provider to supplement registration data. Near the estimated date of delivery, the Registry prompts the health care provider to provide pregnancy outcome data. The data elements requested include:

* Health care provider contact information
* Eligibility criteria
* Uterine fibroid treatment (30 days prior to conception and during pregnancy and includes non-steroidal anti-inflammatory drugs, oral contraceptive pills, progestational agents, gonadotropin-releasing hormone (GnRH) agonists, and other oral agents)
* Pregnancy/Birth outcome
* Maternal information
* Prenatal tests
* Uterine fibroid classification

If a live birth is reported, the Registry conducts the follow-up with the infant's health care provider within 2 months of birth, and at 12 months of age. If a birth defect is indicated, the Registry will request additional targeted follow-up information from the health care provider. Data on any adverse event will be forwarded to the Sponsors.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently pregnant or report is a retrospective defect
* Patient was diagnosed with uterine fibroids prior to becoming pregnant
* Patient is between the ages of 20 and 55

Ages: 20 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2360
Dates: Start 2005-12; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Susan S Roberts, PhD, Study Director — Syneos Health